CLINICAL TRIAL: NCT04720430
Title: Circulating MicroRNA Levels as a Predictor of Successful Bridging or Down-Staging Loco-Regional Therapy (LRT) to Liver Transplantation for Patients With Hepatocellular Carcinoma (HCC)
Brief Title: Blood Sample Collection for Experimental Blood Test to Track Liver Cancer
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 19D.737; JT 13572 (Other: JeffTrial Number)
Record Dates: First submitted 2020-12-07; First posted 2021-01-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study investigates if an experimental blood test can help predict how well cancer will remain under control with treatment. Ther experimental blood test involves measuring mircoRNAs. MicroRNAs are small molecules which help regulate how genes are expressed. This information may help researchers guide treatment for other patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Definite diagnosis of hepatocellular carcinoma established (by standard radiographic or histologic criteria)
* Felt to be reasonable candidate for liver transplantation, potentially contingent on success of down-staging therapy

Exclusion Criteria:

* Either active or recent solid organ cancer other than hepatocellur carcinoma (HCC) within the last 5 years, unless determined by transplant hepatology team not to represent contra-indication to liver transplantation
* Contra-indication to LRT (as assessed by interventional radiologist, for example severe thrombocytopenia, severe vascular disease precluding access, etc)
* History of prior liver transplantation
* Active or prior systemic therapy for HCC

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patientss with hepatocellular carcinoma felt to be reasonable candidate for liver transplantation, potentially contingent on success of down-staging therapy
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Patient Clinical Status - Liver Transplant | At study completion, up to 12 months
  Undergoing liver transplant
Patient Clinical Status - Death | At study completion, up to 12 months
  Will assess the following: death
Patient Clinical Status - Candidacy | At study completion, up to 12 months
  No longer candidate for transplantation for reasons other than tumor progression
Patient Clinical Status | At study completion, up to 12 months
  No longer candidate for transplantation due to tumor progression despite loco-regional therapy efforts
Incidence of "Wait List Drop Off" | At study completion, up to 12 months
  Will be estimated and presented with a Clopper-Pearson exact binomial confidence interval

SECONDARY OUTCOMES:
Time to "Wait List Drop Off" | Up to 12 months
  Cox proportinal hazards modeling will be used to investigate the associations of each micro ribonucleic acid (miRNO) with time to "wait list drop off"
Clinical Status of the subset of patients successfully reaching liver transplant | At 1 year after transplantation
  Logistic regression modeling will be used to investigate the correlation of each miRNA with clincial status (alive without recurrence vs. recurrence or death) within one year of transplant will be cinducted in the subset of those undergoing transplant. The p-values will be adjusted for false discovery rate inflation by the methods of Benjamni & Hochberg (1995) for both secondary analyses, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States